CLINICAL TRIAL: NCT04250818
Title: Predicting Response of Metastatic Triple Negative Breast Cancer to Immunotherapy Based on Patients Cytokine Profile
Status: Suspended | Type: Observational
Why Stopped: PI is moving to a new institution
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Alexander Philipovskiy, Assistant Professor, Texas Tech University Health Sciences Center, El Paso
Other Study IDs: E19137
Record Dates: First submitted 2019-12-18; First posted 2020-01-31 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Triple-Negative Breast Cancer
Keywords: cytokine, breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and whole blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Patients with mTNBC who receive chemotherapy only
- Experimental Group: patients with mTNBC who receive a combination of chemotherapy and Immunotherapy

SUMMARY:
Recent progress in immunotherapy (IT) has shifted treatment paradigms for multiple malignancies including breast cancer. It has been shown that levels of certain cytokines were correlated with increased response to immunotherapy in patients with metastatic breast cancer. In this study investigators will perform cytokine profiling among patients diagnosed with metastatic triple-negative breast cancer at different time points during the treatment.

DETAILED DESCRIPTION:
This is a prospective study that has two groups of patients as determined by their prescribed treatment plan. Group A (control group) are patients with metastatic triple-negative breast cancer (TNBC) who receive chemotherapy only (current standard of care). Group B (experimental group) are patients with mTNBC who receive a combination of chemotherapy and IT immunotherapy (Atezolizumab) which is a standard of care for patients whose tumor express >1% of PD-L1 molecules. T-cell cytokines will be measures prior to treatment and at multiple time points during the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic triple negative breast cancer
* 18 years of age or older

Exclusion Criteria:

* Younger than 18
* Unwilling to participate or unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The majority of the patients with triple negative breast cancer are women
Study Population: Women diagnosed with triple negative breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Tech University HSC El Paso, El Paso, Texas, United States